CLINICAL TRIAL: NCT04760574
Title: Association Between Human Immunodeficiency Virus (HIV) Infection and Male Hypogonadism
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202010105RIND
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Hypogonadism; Ovarian
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: HIV infected men who have sex with men
  Interventions: Diagnostic Test: Testosterone
- Control group: HIV non-infected men
  Interventions: Diagnostic Test: Testosterone

INTERVENTIONS:
Diagnostic Test: Testosterone — Serum total testosterone and free testosterone level

SUMMARY:
Cross-sectional study investigating the prevalence of hypogonadism in HIV-infected MSM population

DETAILED DESCRIPTION:
In this study, we conduct a cross-sectional study investigating the prevalence of hypogonadism in HIV-infected MSM population. Age-matched non-HIV infected MSM group will be used as comparison group. We will also determine the risk factors associated with male hypogonadism (age, duration of HIV infection, comorbidities, BMI, ART use). Correlation will be made between serum testosterone levels and sexual function, vitality, exercise capacity, mood, and bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected men who have sex with men
* HIV non-infected men

Exclusion Criteria:

* Use of testosterone supplement, anabolic steroid in the past one year.
* History of pituitary , adrenal or gonad diseases
* History of pituitary surgery or radiation therapy
* History of systemic chemotherapy
* Active opportunistic infection under treatment
* Cancer
* Severe hepatic, renal or cardiac impairment

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cross-sectional study investigating the prevalence of hypogonadism in HIV-infected MSM population. Age-matched non-HIV infected group will be used as comparison group
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Symptoms of androgen deficiency | 2021-2030
  We use the score of Androgen Deficiency in Aging Males (ADAM) questionnaire to study the prevalence of hypogonadism in HIV-infected MSM population
Serum free testosterone | 2021-2030
  We use serum free testosterone to study the prevalence of hypogonadism in HIV-infected MSM population

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan